CLINICAL TRIAL: NCT01234727
Title: Multicentre Performance Comparison Study of Blood Glucose Monitoring Systems in People With Diabetes Randomised to Multiple Devices
Brief Title: Comparison Study of Blood Glucose Monitoring Systems in People With Diabetes
Status: Completed | Type: Observational
Sponsor: Abbott Diabetes Care (Industry)
Collaborators: ikfe-CRO GmbH (Industry)
Responsible Party: Harald Pohlmeier, Zentrum für Diabetes und Gefäßerkrankungen
Other Study IDs: ADC-MKG-FSL-10008
Record Dates: First submitted 2010-11-03; First posted 2010-11-04 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2011-03

CONDITIONS: Diabetes Mellitus
Keywords: diabetes, SMBG, glucose testing systems, accuracy
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diabetes: Patients with Type 1 or Type 2 diabetes requiring insulin.

SUMMARY:
A Multicentre study comparing 5 different Self-Monitoring Of Blood Glucose (SMBG) system commercially available in Germany & Holland.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with type 1 or type 2 diabetes mellitus
* Age between 18 and 75 years.
* Patients with stable blood glucose in judgment of the investigator.
* Subjects receive intensive insulin therapy (Multiple Daily Injection defined as at least two insulin injections per day)
* Patients perform blood glucose self measurements on a routine basis
* Patients must have experience in self measurement blood glucose for at least 6 months.

Exclusion Criteria:

* Patients with unstable blood glucose in judgment of the investigator.
* Patient has been diagnosed with progressive / serious diseases that in judgment of the investigator preclude successful completion of the observational period.
* Lack of compliance or other justifications that, in the discretion of the investigator, precludes satisfactory participation in the study.
* Subject without legal capacity.
* Blood donation within the last 30 days.
* Known pregnancy.
* Subject has already participated in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 480 subjects with type 1 or 2 diabetes mellitus
Sampling Method: Non-Probability Sample
Enrollment: 501 (Actual)
Dates: Start 2010-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joe Bugler, Study Director — Abbott Diabetes Care
Locations (3):
- Germany (2):
  - Zentrum für Diabetes und Gefäßerkrankungen, Münster
  - Diabetes Zentrum Neuwied, Neuwied
- Radboud University Nijmegen Centre, Nijmegen, Netherlands